CLINICAL TRIAL: NCT03448042
Title: A Phase Ia/Ib, Open-Label, Dose-Escalation Study of the Safety and Pharmacokinetics of Runimotamab Administered Intravenously as a Single Agent and in Combination With Trastuzumab in Patients With Locally Advanced or Metastatic HER2-Expressing Cancers
Brief Title: A Study of Runimotamab in Participants With Locally Advanced or Metastatic HER2-Expressing Cancers
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GO40311
Record Dates: First submitted 2018-02-20; First posted 2018-02-27 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Solid Tumors
MeSH Terms: interventions — Trastuzumab; tocilizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation (Experimental): Participants will be assigned sequentially to escalating doses of runimotamab up to the maximum tolerated dose (MTD).
  Interventions: Drug: Runimotamab; Drug: Trastuzumab; Drug: Tocilizumab
- Dose Expansion (Experimental): Participants will receive runimotamab based on the MTD or maximum allowed dose (MAD) identified during dose escalation.
  Interventions: Drug: Runimotamab; Drug: Trastuzumab; Drug: Tocilizumab

INTERVENTIONS:
Drug: Runimotamab — Runimotamab will be administered via IV infusion until disease progression, intolerable toxicity, or any other discontinuation criteria are met.
  Other Names: BTRC4017A; RO7227780
Drug: Trastuzumab — Trastuzumab will be administered via IV infusion
Drug: Tocilizumab — Participants will receive IV tocilizumab if needed

SUMMARY:
This study will evaluate the safety, tolerability, and pharmacokinetics of Runimotamab administered intravenously as a single agent and in combination with Trastuzumab in participants with locally advanced or metastatic Human Epidermal Growth Factor Receptor 2 (HER2)-expressing cancers.

ELIGIBILITY:
Inclusion Criteria

* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Life expectancy of at least 12 weeks
* Adequate hematologic and end-organ function
* Acute, clinically significant treatment-related toxicity from prior therapy must have resolved to Grade </=1 prior to study entry
* Left Ventricular Ejection Fraction (LVEF) >/=50%

HER2-Expressing Breast Cancer-Specific Inclusion Criteria

* Locally tested, Human Epidermal Growth Factor Receptor 2 (HER2)-expressing BC
* Locally advanced or metastatic BC that has relapsed or is refractory to established therapies

HER2-Expressing Gastric/Gastroesophageal (GEJ) Cancer-Specific Inclusion Criteria

* Adenocarcinoma of the stomach or GEJ with inoperable locally advanced or recurrent and/or metastatic disease, not amenable to curative therapy
* HER2-expressing tumor (primary tumor or metastasis) as assessed by local lab testing
* HER2-positive gastric/GEJ cancer must have received prior trastuzumab, cisplatin (or carboplatin or oxaliplatin or investigational platinum agent) and 5-fluorouracil (5-FU)/capecitabine

HER2-Positive Solid Tumor Specific Inclusion Criteria

* HER2-positive tumor (primary tumor or metastasis) as assessed by local (non-central) laboratory testing
* Locally advanced, recurrent, or metastatic incurable malignancy that has progressed after at least one available standard therapy; or for whom standard therapy has proven to be ineffective or intolerable, or is considered inappropriate; or for whom a clinical trial of an investigational agent is a recognized standard of care; or for whom a clinical trial of an investigational agent is considered an acceptable treatment option

Exclusion Criteria

* Pregnant or breastfeeding, or intending to become pregnant during the study or within 140 days after the last dose of runimotamab
* Significant cardiopulmonary dysfunction
* Known clinically significant liver disease
* Positive for acute or chronic Hepatitis B virus (HBV) infection
* Acute or chronic Hepatitis C virus (HCV) infection
* Human Immunodeficiency Virus (HIV) seropositivity
* Poorly controlled Type 2 diabetes mellitus
* History of ventricular dysrhythmias or risk factors for ventricular dysrhythmias
* Current treatment with medications that are well known to prolong the Q-wave/T-wave (QT) interval
* Known clinically significant liver disease
* Primary central nervous system (CNS) malignancy, untreated CNS metastases, or active CNS metastases (progressing or requiring corticosteroids for symptomatic control)
* Leptomeningeal disease
* Spinal cord compression that has not definitively treated with surgery and/or radiation
* History of autoimmune disease
* Prior allogeneic stem cell or solid organ transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2018-06-06 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Adverse Events | From baseline through end of study (approximately 78 months)

SECONDARY OUTCOMES:
Serum Concentration of Runimotamab | At predefined intervals from Cycle 1, Day 1 (approximately 1 year)
Area Under the Serum Concentration vs. Time Curve (AUC) of Runimotamab | At predefined intervals from Cycle 1, Day 1 (approximately 1 year)
Maximum Observed Serum Concentration (Cmax) of Runimotamab | At predefined intervals from Cycle 1, Day 1 (approximately 1 year)
Minimum Observed Serum Concentration (Cmin) of Runimotamab | At predefined intervals from Cycle 1, Day 1 (approximately 1 year)
Clearance (CL) of Runimotamab | At predefined intervals from Cycle 1, Day 1 (approximately 1 year)
Volume of Distribution at Steady State (Vss) of Runimotamab | At predefined intervals from Cycle 1, Day 1 (approximately 1 year)
Objective Response (OR) as Determined by the Investigator According to Response Evaluation Criteria In Solid Tumors v1.1 (RECIST v1.1) | Baseline through the end of study (approximately 78 months)
Duration of Response (DOR) | From the first occurrence of a documented objective response to first documented disease progression or death from any cause, through the end of the study (approximately 78 months)
Anti-Drug Antibody (ADA) Levels of Runimotamab | At predefined intervals from Cycle 1, Day 1 (approximately 1 year)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (27):
- United States (5):
  - Yale University, New Haven, Connecticut
  - Washington University, Saint Louis, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - SCRI Oncology Partners, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
- Peter MacCallum Cancer Centre, Melbourne, Victoria, Australia
- Grand Hopital de Charleroi asbl, Charleroi, Belgium
- Princess Margaret Hospital, Toronto, Ontario, Canada
- Rigshospitalet-Blegdamsvej 9, Copenhagen, Denmark
- France (4):
  - EDOG - Institut Bergonie - PPDS, Bordeaux, Gironde
  - Centre Léon Bérard, Lyon, Rhône
  - Gustave Roussy, Villejuif, Val-de-Marne
  - Institut Claudius Regaud, Toulouse
- ASST Grande Ospedale Metropolitano Niguarda - Presidio Ospedaliero Ospedale Niguarda Ca' Granda, Milan, Lombardy, Italy
- National Cancer Center East, Chiba, Japan
- Het Nederlands Kanker Instituut Antoni Van Leeuwenhoek Ziekenhuis, Amsterdam, Netherlands
- National Cancer Centre, Singapore, Singapore
- South Korea (2):
  - Asan Medical Center, Seoul
  - Seoul National University Hospital, Seoul
- Spain (5):
  - Hospital Universitario Quironsalud Madrid, Pozuelo de Alarcón, Madrid
  - Hospital Universitari Vall d'Hebron, Barcelona
  - START MADRID_Hospital Universiario Fundacion Jimenez Diaz, Madrid
  - START MADRID_Hospital Universitario HM Sanchinarro - CIOCC - EDOS, Madrid
  - Hospital Clinico Universitario de Valencia, Valencia
- Taiwan (2):
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
- Churchill Hospital, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No